CLINICAL TRIAL: NCT00359112
Title: A Randomised, Multi-Centre, Phase IV, Double-Blind, Parallel Group Study Comparing the Effects of 52 Weeks Administration of AVANDAMET and Metformin Plus Sulphonylurea on Change in HbA1c From Baseline in Overweight Type 2 Diabetics Poorly Controlled on Metformin.
Brief Title: AVANDAMET Versus Metformin And Sulphonylurea In People With Poorly Controlled Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVM100264
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-05

CONDITIONS: Non-Insulin-Dependent Diabetes Mellitus
Keywords: Type 2 diabetes; overweight; AVANDAMET; metformin; sulphonylurea
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight | interventions — Metformin; Sulfonylurea Compounds; rosiglitazone-metformin combination

INTERVENTIONS:
Drug: metformin
Drug: sulphonylurea
Drug: Avandamet
  Other Names: metformin; sulphonylurea

SUMMARY:
This study compares the effects of Avandamet (rosiglitazone maleate/metformin) treatment and metformin plus sulphonylurea treatment in overweight people with type 2 diabetes.

ELIGIBILITY:
Inclusion criteria:

* Body mass index > or = to 25 kg/m2.
* HbA1c > or =7% and < or =10% at screening.
* FPG > or = 7.0mmol/L (126mg/dL) at visit 2.
* Receiving at least 0.85g of metformin at constant dose(s) for at least 8 weeks prior to visit 1a.
* Female subjects must be postmenopausal or using effective contraceptive measures.

Exclusion criteria:

* Use of any other oral antidiabetic drug other than metformin within 12 weeks prior to screening.
* Subjects with clinically significant ongoing oedema requiring pharmacological treatment or with a history of oedema requiring pharmacological treatment.
* Subjects with a history of severe hypoglycaemia.
* Renal disease or renal dysfunction.
* Presence of clinically significant hepatic disease.
* Presence of unstable or severe angina or known NYHA grade I-IV congestive heart failure.
* Subjects who have had a previous myocardial infarction, percutaneous transluminal coronary angioplasty, coronary artery bypass graft or cerebrovascular accident within 3 months prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 544
Dates: Start 2004-02

PRIMARY OUTCOMES:
Change in HbA1c level from baseline following 52 weeks of treatment.

SECONDARY OUTCOMES:
Change in FPG (fasting plasma glucose)
insulin sensitivity
beta cell function
change in PAI-1
CRP
number of hypoglycaemic events
Change in 24 hr ABPM
Diabetes treatment satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, DM, FRCP, Study Director — GlaxoSmithKline
Locations (130):
- Belgium (11):
  - GSK Investigational Site, Bruges
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Champion
  - GSK Investigational Site, Heverlee
  - GSK Investigational Site, Landen
  - GSK Investigational Site, Oostham
  - GSK Investigational Site, Petit-Rechain
  - GSK Investigational Site, Pulle
  - GSK Investigational Site, Tessenderlo
  - GSK Investigational Site, Tremelo
  - GSK Investigational Site, Willebroek
- France (15):
  - GSK Investigational Site, Roubaix, Hauts-de-France
  - GSK Investigational Site, Anzin
  - GSK Investigational Site, Briollay
  - GSK Investigational Site, Commelle
  - GSK Investigational Site, Cremeaux
  - GSK Investigational Site, Évron
  - GSK Investigational Site, Laval
  - GSK Investigational Site, Louverné
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Roanne
  - GSK Investigational Site, Saint-Ouen
  - GSK Investigational Site, Sainte-Suzanne
  - GSK Investigational Site, Segré
  - GSK Investigational Site, Vénissieux
- Germany (34):
  - GSK Investigational Site, Güglingen, Baden-Wurttemberg
  - GSK Investigational Site, Kippenheim, Baden-Wurttemberg
  - GSK Investigational Site, Königsfeld im Schwarzwald, Baden-Wurttemberg
  - GSK Investigational Site, Waldshut-Tiengen, Baden-Wurttemberg
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Grafing, Bavaria
  - GSK Investigational Site, Herzogenaurach, Bavaria
  - GSK Investigational Site, Immenstadt im Allgäu, Bavaria
  - GSK Investigational Site, Oberteisendorf, Bavaria
  - GSK Investigational Site, Saaldorf, Bavaria
  - GSK Investigational Site, Wallerfing, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Großalmerode, Hesse
  - GSK Investigational Site, Einbeck, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Isernhagen-Süd, Lower Saxony
  - GSK Investigational Site, Papenburg, Lower Saxony
  - GSK Investigational Site, Beckum, North Rhine-Westphalia
  - GSK Investigational Site, Bergkamen-Rünthe, North Rhine-Westphalia
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Dinslaken, North Rhine-Westphalia
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Viersen, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Neuwied, Rhineland-Palatinate
  - GSK Investigational Site, Rhaunen, Rhineland-Palatinate
  - GSK Investigational Site, Speyer, Rhineland-Palatinate
  - GSK Investigational Site, Saarlouis, Saarland
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Wolmirstedt, Saxony-Anhalt
  - GSK Investigational Site, Elmshorn, Schleswig-Holstein
- Ireland (2):
  - GSK Investigational Site, Blanchardstown
  - GSK Investigational Site, Dublin
- Italy (8):
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Ferrara, Emilia-Romagna
  - GSK Investigational Site, Ravenna, Emilia-Romagna
  - GSK Investigational Site, Arenzano (GE), Liguria
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Sassari, Sardinia
  - GSK Investigational Site, Città Di Castello (PG), Umbria
  - GSK Investigational Site, Terni, Umbria
- Lithuania (2):
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Vilnius
- Mexico (5):
  - GSK Investigational Site, Tijuana, Baja California Norte
  - GSK Investigational Site, Durango, Durango
  - GSK Investigational Site, Pachuca, Hidalgo
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Mexico City
- Netherlands (12):
  - GSK Investigational Site, Beek en Donk
  - GSK Investigational Site, Beerzerveld
  - GSK Investigational Site, Heerlen
  - GSK Investigational Site, Hoogvliet
  - GSK Investigational Site, Landgraaf
  - GSK Investigational Site, Musselkanaal
  - GSK Investigational Site, Oude Pekela
  - GSK Investigational Site, Spijkenisse
  - GSK Investigational Site, The Hague
  - GSK Investigational Site, Woerden
  - GSK Investigational Site, Zaandam
  - GSK Investigational Site, Zieuwent
- Spain (23):
  - GSK Investigational Site, Alcobendas/Madrid
  - GSK Investigational Site, Alcora/Castellón
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Alzira
  - GSK Investigational Site, Artana/Castellón
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Benicassim (Castellon)
  - GSK Investigational Site, Cadiz
  - GSK Investigational Site, Castellon
  - GSK Investigational Site, Cáceres
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Mérida
  - GSK Investigational Site, Móstoles/Madrid
  - GSK Investigational Site, Onda (Castellon)
  - GSK Investigational Site, Pontevedra
  - GSK Investigational Site, Sabadell (Barcelona)
  - GSK Investigational Site, Sant Joan d'Alacant
  - GSK Investigational Site, Santa Coloma de Gramanet (Barcelona)
  - GSK Investigational Site, Tarrasa, Barcelona
  - GSK Investigational Site, Valencia
- Switzerland (12):
  - GSK Investigational Site, Bern
  - GSK Investigational Site, Emmenbrücke
  - GSK Investigational Site, Gettnau
  - GSK Investigational Site, Jegenstorf
  - GSK Investigational Site, Lucerne
  - GSK Investigational Site, Lugano
  - GSK Investigational Site, Pregassona
  - GSK Investigational Site, Salmsach
  - GSK Investigational Site, St-Maurice
  - GSK Investigational Site, Steckborn
  - GSK Investigational Site, Winterthur
  - GSK Investigational Site, Zurich
- United Kingdom (6):
  - GSK Investigational Site, Glasgow, Lanarkshire
  - GSK Investigational Site, Blackpool, Lancashire
  - GSK Investigational Site, Bath, Somerset
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, Sheffield